CLINICAL TRIAL: NCT05541159
Title: A Phase 1, Open-label, Single-dose, Multi-center, Parallel Group Study to Evaluate the Pharmacokinetics of TNO155 in Participants With Mild, Moderate, or Severe Renal Impairment Compared to Matched Healthy Control Participants
Brief Title: Pharmacokinetics Study of TNO155 in Participants With Mild, Moderate, or Severe Renal Impairment Compared to Matched Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTNO155A12105
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Renal Impairment
Keywords: TNO155; renal Impairment; SHP2
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: The study will be divided into 2 parts. Participants in the renal impairment groups will be staged by their respective degree of renal function (mild, moderate, or severe) according to the estimated glomerular filtration rate determined at the screening visit.
  Healthy participants who were identified and enrolled as matching partners for a renal impairment group in Part I can serve as matching partners for participants in renal impairment group (Group 4) in Part II if they fulfilled the matching criteria. Otherwise, additional matched healthy participants will be enrolled.
  Part I: will include participants with mild and moderate levels of renal impairment as well as healthy control participants Part II: will include participants with severe renal impairment, if allowed after results of interim analysis (IA) obtained for mild and moderate groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Healthy control participants with normal renal function
  Interventions: Drug: TNO155
- Group 2 (Experimental): Mild renal impairment
  Interventions: Drug: TNO155
- Group 3 (Experimental): Moderate renal impairment
  Interventions: Drug: TNO155
- Group 4 (Experimental): Severe renal impairment
  Interventions: Drug: TNO155

INTERVENTIONS:
Drug: TNO155 — Single oral dose of TNO155 on Day 1

SUMMARY:
The purpose of this Phase 1 study is to evaluate the effect of various degrees of renal impairment on plasma pharmacokinetics (PK), safety and tolerability of TNO155. The results of this study will guide the Novartis recommendation regarding whether or not a dose adjustment may be needed when treating patients with renal impairment

DETAILED DESCRIPTION:
This is a study to evaluate the PK of TNO155 in participants with mild, moderate or severe renal impairment compared to matched healthy control participants with normal renal function. The study will be divided into 2 parts. Participants in the renal impairment groups will be staged by their respective degree of renal function (mild, moderate, or severe) according to the estimated glomerular filtration rate (eGFR) determined at the screening visit. Each renal impairment participant must be matched to a healthy control participant with respect to age (±10 years), body weight (±20%) and sex. Each participant in the healthy control group (Group 1) can be matched to one or more participants from any renal impairment group (Groups 2, 3, and 4).

On Day 1 morning, participants will receive a single oral dose of TNO155 .All participants will be domiciled from Day -1 until Day 11. All participants should have a poststudy safety follow-up contact conducted approximately 30 days after administration of study treatment. The study will be considered complete once all the participants have finished the required assessments, dropped out, or been lost to follow-up before completing the required assessments.

ELIGIBILITY:
Inclusion Criteria:

All participants Participants must weigh at least 50 kg and no more than 120 kg and must have a body mass index (BMI) within the range of 18.0 to 38.0 kg/m2, inclusive, for healthy participants. Must be a non-smoker or and agree to remain a non-smoker from screening until the End of Study.

Group 1

•eGFR as determined by Chronic Kidney Disease Epidemiology Collaboration [CKD EPI] equation and conversion within normal range as determined by GFR 90 mL/min at screening and baseline.

Groups 2 to 4

* Participants with different levels of impaired renal function satisfying criteria for renal impairment as determined at screening by the eGFR at screening
* Participants must have documented stable renal disease without evidence of renal progressive disease

Exclusion Criteria:

All Participants

* Use of drugs (prescription, non-prescription and herbal remedies such as St John's wort), within 4 weeks prior to dosing until completion of the End of Study Visit.
* Participant has received a renal transplant at any time in the past and is on immunosuppressant therapy Left ventricular ejection fraction (LVEF) < 50% or below the institutional standard lower limit, at screening or baseline.
* Uncontrolled hypertension despite medical treatment at screening or baseline. Group 1
* Significant illness, which has not been resolved within 2 weeks prior to dosing of study treatment.
* History or presence of renal disease or kidney injury Groups 2, 3 and 4
* Severe albuminuria
* Other laboratory values grade 2 severity according to NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE)
* Participants undergoing any method of dialysis.
* Participants with renal impairment due to hepatic disease (hepatorenal syndrome).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-19 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-versus-time curve (AUC) from time zero to the last measurable plasma concentration (AUClast) of TNO155 | Up to 240 hours post single dose
  AUClast will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
AUC from time zero to time "t" (AUC0-t) of TNO155 | AUC from time zero to time "t" (AUC0-t) of TNO155
  AUC0-t will be calculated as needed based on TNO155 plasma concentrations and non-compartmental methods. The definition of time "t" may be data-driven post-hoc to mitigate treatment bias due to within participant differences in Tlast between the treatments, or may be selected to allow between-study exposure comparisons that use a common time window.
AUC from time zero to infinity (AUCinf) of TNO155 | Up to 240 hours post single dose
  AUCinf will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Maximum (peak) observed plasma concentration (Cmax) of TNO155 | Up to 240 hours post single dose
  Cmax will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Time to reach maximum observed plasma concentration (Tmax) of TNO155 | Up to 240 hours post single dose
  Tmax will be calculated based on TNO155 plasma concentrations and non-compartmental methods
Elimination half-life (T1/2) of TNO155 | Up to 240 hours post single dose
  T1/2 will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Sampling time of the last measurable plasma concentration (Tlast) of TNO155 | Up to 240 hours post single dose
  Tlast will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Apparent plasma clearance (CL/F) of TNO155 | Up to 240 hours post single dose
  CL/F will be calculated based on TNO155 plasma concentrations and non-compartmental methods.
Apparent volume of distribution during terminal phase (Vz/F) of TNO155 | Up to 240 hours post single dose
  Vz/F will be calculated based on TNO155 plasma concentrations and non-compartmental methods.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days post single dose
  Incidence of AEs and SAEs, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Unbound Cmax (Cmax,u) of TNO155 | Up to 240 hours post single dose
  Cmax,u will be calculated based on the unbound fraction of TNO155 in plasma.
Unbound AUClast (AUClast,u) of TNO155 | Up to 240 hours post single dose
  AUClast,u will be calculated based on the unbound fraction of TNO155 in plasma.
Unbound AUCinf (AUCinf,u) of TNO155 | Up to 240 hours post single dose
  AUCinf,u will be calculated based on the unbound fraction of TNO155 in plasma
Unbound CL/F (CL/F,u) of TNO155 | Up to 240 hours post single dose
  CL/F,u will be calculated based on the unbound fraction of TNO155 in plasma.
Renal clearance (CLr) of TNO155 | Up to 240 hours post single dose
  CLr will be calculated based on urinary excretion data of TNO155.
Apparent non-renal clearance (CLNR/F) of TNO155 | Up to 240 hours post single dose
  CLNR/F will be calculated based on urinary excretion data of TNO155.
Fraction of dose excreted in urine (fe) of TNO155 | Up to 240 hours post single dose
  Fe will be calculated based on urinary excretion data of TNO155.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No